CLINICAL TRIAL: NCT06218160
Title: A Randomized Controlled Study of Ropivacaine Combined With Hydromorphone to Block Lumbar Muscle in Elderly Inguinal Hernia Repair.
Brief Title: The Addition of Hydromorphone to Local Anesthetics for the Repair of Inguinal Hernias in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/148
Record Dates: First submitted 2023-12-30; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Inguinal Hernia
Keywords: hydromorphone; Quadratus lumbois block; old people
MeSH Terms: conditions — Hernia, Inguinal | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydromorphone combined with ropivacaine (Experimental): The posterior quadrat block was performed by adding 1mg hydromorphone to 0.375% ropivacaine in a total of 30ml.
  Interventions: Drug: Hydromorphone combined with ropivacaine
- ropivacaine (Active Comparator): A mixture of 0.375% ropivacaine for a total of 30ml was performed for posterior quadrate block.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Hydromorphone combined with ropivacaine — 1mg hydromorphone was added to 0.375% ropivacaine for a total of 30ml to perform quadrat block
  Other Names: Quadratus lumbois block
  Arms: Hydromorphone combined with ropivacaine
Drug: Ropivacaine — A mixture of 0.375% ropivacaine for a total of 30ml was used for quadrate block
  Other Names: Quadratus lumbois block
  Arms: ropivacaine

SUMMARY:
To compare the clinical and postoperative analgesic effects of hydromorphone combined with ropivacaine and ropivacaine alone in quadrangular muscle block for open inguinal hernia in elderly patients.

DETAILED DESCRIPTION:
Elderly patients selected for Lichtenstein hernia repair in our hospital who met the inclusion and exclusion criteria and obtained informed consent were included in this trial, and were randomly divided into experimental group by random number table method: 0.375% ropivacaine combined with hydromorphone block group, and control group: 0.375% ropivacaine block group alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and above.
* Admission to hospital for open inguinal hernia surgery is consistent with the -indications of this surgical modality, ASA grades 1 to 3.
* No recent use of sedatives, opioids, or other analgesics.
* Good compliance, signed informed consent.
* Complete clinical data.

Exclusion Criteria:

* There are serious cardiovascular and cerebrovascular diseases.
* Abdominal infection.
* Coagulation dysfunction or receiving anticoagulation therapy.
* Local anesthesia drug allergy.
* Can not cooperate with the corresponding operation, suffering from mental illness.
* Previous surgical history of the corresponding position in the abdomen that may interfere with the surgical process of this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Related indexes of anesthesia effect: pain after surgery, 6, 12, 18,24, 48h after surgery. | From the end of surgery until two days after surgery.
  Visual analogue scale (VAS) was used to score the postoperative pain at 6,12,18,24,48h.The score ranges from 0 (no pain) to 10 (most severe pain). The change was equal to the score difference between the two groups at different observation time points (6,12,18,24,48h).
Related indexes of anesthesia effect: time of onset of anesthesia, duration of anesthesia maintenance. | From the start of anesthesia until two days after surgery.
  The range of the effective time of anesthesia minus the start time of anesthesia and the maintenance time minus the start time of anesthesia are respectively.The unit of time is minutes.

SECONDARY OUTCOMES:
The occurrence of postoperative adverse reactions. | The operation ended two days after surgery.
  The rates of postoperative nausea, vomiting and dizziness were compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Tian, Study Director — Second Hospital of Jilin University
Locations (1):
- Second Hospital of Jilin University, Changchun, Jilin, China